CLINICAL TRIAL: NCT02575560
Title: High Dose Weekly Use First-generation EGFR-TKI Instead of Daily Regular Dose in the Treatment of EGFR-TKI Acquired Resistance Non-small Cell Lung Cancer (NSCLC)
Brief Title: Weekly Use First-generation EGFR-TKI in the Treatment of EGFR-TKI Acquired Resistance Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, Director, Qingdao Central Hospital
Other Study IDs: QCH200501
Record Dates: First submitted 2015-10-08; First posted 2015-10-14 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2015-10

CONDITIONS: EGFR-TKI Resistant Mutation
Keywords: Progression-Free Survival

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- weekly use erolotinib vs history data: Drug: erolotinib erolotinib 1050mg, oral, once a week, continues to disease progression or death or stop by physician
  Interventions: Other: history data

INTERVENTIONS:
Other: history data — history data of PFS after 1st line or second line theray

SUMMARY:
EGFR-TKI is the main is the first line therapy for local advanced or metastatic non-small cell lung cancer with EGFR gene mutation. The median progression free survival time is around 11 months with the first generation EGFR-TKI. Patients with acquired resistance with first generation EGFR-TKI usually with EGFR exon 20 mutation (T790M). Change the drug administration maybe prolong patients PFS and evently prolong OS.

DETAILED DESCRIPTION:
1st generation EGFR-TKI has reversible binding to EGFR, it also bind to T790M in a high dose which is account about 60% patients acquired resistance to the drug. Resistance patients may be benefit to a bolus drug use to block T790M gene.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC with EGFR mutation progressed after first generation EGFR-TKI, or progressed after chemotherapy and 1st generation EGFR-TKI or progressed after 1st generation EGFR-TKI and chemotherapy. Expected survival more than 3 months with a ECOG ≤3.

Exclusion Criteria:

* liver function (ALT, AST) and renal function 2 times higher than normal limit; IPD; uncontrolled diarrhea; severe anemia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: histological confirmed local advanced or metastatic lung adenocarcinoma with EGFR mutation diagnosed by 2nd generation sequence system.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10-01; Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival Time (PFS) | an average 1 year

SECONDARY OUTCOMES:
Overall Response Rate(ORR) | an average half year
Overall Survival Time (OS) | an average 2 year

CONTACTS AND LOCATIONS:
Overall Officials: ketao lan, Study Chair — Qingdao Central Hospital
Locations (1):
- Qingdao Central Hospital, Qingdao, Shandong, China